CLINICAL TRIAL: NCT00292734
Title: Additive Beneficial Effect of Zolpidem Onto the Antidepressant Therapy in Depressive and Dysthimic Patients in the Acute Phase of the Disease
Brief Title: STILDEP: Zolpidem in Depressive and Dysthimic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: L_9259; EudraCT # : 2004-001967-24
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Sleep Initiation and Maintenance Disorders; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Zolpidem

INTERVENTIONS:
Drug: Zolpidem

SUMMARY:
Primary objective: To show that the combination of Zolpidem + antidepressant therapy is more effective in the treatment of the secondary insomnia of depressive and dysthimic patients than antidepressant therapy alone in the acute phase of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Depressive and dysthimic patients in acute phase of mild to moderate severity
* Depressive and dysthimic patients suffering from secondary insomnia (DSM IV) recent antidepressant therapy (less than 1 week)

Exclusion Criteria:

* Regularly use of sleeping pills in the last 2-3 month
* Use of any sleeping pils in the last week
* Insufficient hepatic
* Myasthenia gravis
* Proven hypersensivity to Zolpidem
* Evidence of clinically relevant nervous system disorders (other neurologic/psychiatric diseases associated with depression)
* History of evidence of alcohol or drug abuse
* Evidence of clinically relevant cardiovascular, haematologic, hepatic, gastrointestinal, renal, pulmonary or endocrinologic diseases
* Abnormal snore
* Work an alternating shift
* Suffering from periodic leg movement disorder and sleep apnea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-01; Study Completion 2006-06

PRIMARY OUTCOMES:
To show that the combination of Stilnox+ antidepressant therapy is more effective in the treatment of the secondary insomnia of depressive and dysthimic patients than antidepressant therapy alone in the acute phase of the disease

CONTACTS AND LOCATIONS:
Overall Officials: László Erős, MD, Study Director — sanofi-aventis Hungary
Locations (1):
- Sanofi-Aventis, Budapest, Hungary